CLINICAL TRIAL: NCT03929172
Title: A First-in-Human, Phase 1, Randomized, Placebo-Controlled, Double-Blind Study to Assess the Safety and Tolerability, and to Explore Immunological Effects of I.M. Administered AAVLP-HPV Vaccine in Healthy Adult Male and Female Subjects
Brief Title: A Study of Safety, Tolerability and Immunogenicity of HPV-L2 Vaccine in Healthy Adult Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 2A Pharma AB (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2AP01-01; 2018-003045-42 (EudraCT Number)
Record Dates: First submitted 2019-04-12; First posted 2019-04-26 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Papillomavirus Infections
Keywords: HPV-L2
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAVLP-HPV Vaccine Arm (Experimental): Subjects will receive a total of 3 vaccinations: a prime on Day 1, and boosts on Day 57 (± 2 days) and Day 180 (± 1 week).
  Interventions: Biological: AAVLP-HPV
- Placebo Arm (Placebo Comparator): Subjects will receive a total of 3 vaccinations: a prime on Day 1, and boosts on Day 57 (± 2 days) and Day 180 (± 1 week).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AAVLP-HPV — 20μg/injection formulated in a ready to use solution containing 100mM sodium citrate, 2.5 mM MgCl2, 0.001% pluronic F-68, pH 6.0 for i.m. injection as 0.5 mL per injection.
  Other Names: 2AP01
  Arms: AAVLP-HPV Vaccine Arm
Drug: Placebo — 0.5 mL 100 mM Sodium Citrate, 2.5 mM MgCl2, 0.001% Pluronic F-68, pH 6 for i.m. injection as 0.5 mL per injection.
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and the immunological effects of adeno-associated virus-like particle human papillomavirus (AAVLP-HPV) vaccine in healthy adults.

DETAILED DESCRIPTION:
2A Pharma's AAVLP-HPV vaccine candidate is based on AAVLPs with insertion of sequences of the L2 minor HPV capsid protein. The vaccine's intended clinical use is as a vaccine for prophylaxis against HPV infection in adolescents and adults.

This is a 12 month single-center, randomized, placebo-controlled, double-blind, repeated dose, safety, tolerability, and immunological effect study. Twenty (20) healthy, adult male and female subjects will be enrolled with a minimum of 40% of each gender. Sixteen (16) subjects will be randomized to receive the active drug and 4 subjects to receive the placebo. At least 1 subject of each gender will be randomized to receive the placebo.

Subjects will receive a total of 3 doses of AAVLP-HPV or placebo: a prime on Day 1, and two boosts, one on Day 57 (±2 days) and one on Day 180 (±1 week). The volunteers will be followed until day 365 (±1 week) when they return for the final safety and serum-based immunogenicity and neutralising antibodies assessment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study:

1. Healthy, adult, male or female aged between 18 and 45 years, inclusive, at screening.
2. Body Mass Index (BMI) ≥ 18 and ≤ 32.0 kg/m2 at screening.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
4. For a female of childbearing potential: either be sexually inactive (abstinent as a lifestyle*) for 28 days prior to the first dosing and throughout the study or be using one of the following acceptable birth control methods:

   * hormonal oral contraceptives, vaginal ring, transdermal patch, or hormone releasing intrauterine device for at least 3 months prior to the first dosing with either a physical (e.g., condom, diaphragm, or other) or a chemical (e.g., spermicide) barrier method from the time of screening and throughout the study.
   * depot/implantable hormone (e.g., Depo-provera®, Implanon) for at least 3 months prior to the first dosing and throughout the study.

   In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for at least 28 days following the last dose.

   * True abstinence is defined as refraining from heterosexual intercourse in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to study drug, and withdrawal are not acceptable methods of contraception.
5. For a female of non-childbearing potential: must have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
6. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

Subjects must not be enrolled in the study if they meet any of the following criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
6. Prior vaccination against HPV.
7. Positive for HPV antibodies against HPV types 6, 11, 16, and 18.
8. Have received an investigational vaccination within 90 days before screening.
9. Have received any licensed vaccination within 30 days before screening.
10. Any condition that may interfere with the intended administration of the study drug.
11. Suffered from febrile or infectious illness within 7 days prior to Day 1.
12. Subjects who plan to become pregnant/start a family during the study.
13. Female subjects with a positive pregnancy test or who are lactating.
14. Drink alcohol in excess of 21 glasses/units (425 g) per week for males or 14 glasses/units (284 g) per week for females, with one unit = 150 mL of wine or 360 mL of beer or 45 mL of 45% alcohol.
15. Positive urine drug or alcohol results at screening or Day -1.
16. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
17. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
18. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
19. QTcF interval is >460 msec (males) or >470 msec (females) or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening.
20. Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements that could adversely affect the immune system during 3 months prior to vaccination and throughout the study. Inhaled and topical corticosteroids will be allowed. Medication listed as part of acceptable birth control methods and hormone replacement therapy will be allowed. After randomization, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee. Appropriate sources will be consulted by the PI or designee to confirm interaction with study drugs. Subjects may not initiate new prescription medication within 1 month prior to screening, with exceptions, or must be on a stable dose for at least 90 days prior to vaccination as approved in advance by the PI or designee.
21. Donation of blood or plasma within 90 days prior to the first dosing.
22. Donation of bone marrow within the last 6 months prior to the first dosing.
23. Participation in another clinical study with an investigational agent within the 90 days prior to first dosing. The 90-day window will be derived from the date of the last dosing, whichever is later, in the previous study to Day 1 of the current study.
24. Has tattoo(s) or scarring at or near the site of vaccine administration or any other condition which may interfere with injection site examination, in the opinion of the PI.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects Reporting Solicited Local Symptoms | Day 0 and 1 after each vaccination
  Solicited local symptoms assessed including pain, tenderness, redness, swelling, and induration.
Percentage of Subjects Reporting Solicited General Symptoms | Through 365 days
  Solicited general symptoms assessed including fever, headache, fatigue, nausea, diarrhea, vomiting, myalgia, allergic reaction.
Percentage of Subjects Reporting Unsolicited Adverse Events (AEs) | Through 365 days
  An unsolicited adverse event is defined as any adverse event (AE) reported in addition to those solicited during the clinical study.
Percentage of Subjects Reporting New Onset of Chronic Illness (NOCI) | Through 365 days
  A NOCI is defined as diagnosis post study drug administration of a new medical condition, which is chronic in nature, including those potentially controllable by medication (e.g., diabetes, asthma)
Percentage of Subjects Reporting Adverse Events of Special Interest (AESI) | Through 365 days
  An AESI should not necessarily be classified to be a serious adverse event, even though the event may be clinically significant. If an AESI is reported, the Sponsor should be promptly informed and information relevant to the event should be promptly collected using the same process as that used for reporting serious adverse events. For this protocol, AESI includes demyelinating syndromes or neurological conditions such as complex regional pain or postural orthostatic tachycardia syndromes.
Percentage of Subjects Reporting Serious Adverse Events (SAEs) | Through 365 days
  SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Vital Signs - Body Temperature | Through 365 days
  Single measurements of body temperature 35.6 ≤ Temperature ≤37.7 (C)
Vital Signs - Respiratory Rate | Through 365 days
  Measurements of respiratory rate 8≤ Respiration ≤24 (breaths/min)
Vital Signs - Blood Pressure | Through 365 days
  Measurements of blood pressure 90≤ Systolic ≤140 (mmHg) and 40≤ Diastolic ≤90 (mmHg
Vital Signs - Heart Rate | Through 365 days
  Measurements of 40≤ Pulse ≤99 (beats/min)
Vital Signs - Body Mass Index (BMI | Through 365 days
  Calculated as weight in kg / height in meters^2
Electrocardiogram (ECG) | Through 365 days
  Single 12-lead ECGs will be performed. Measurement type must be one of the following: HR (50≤HR≤100 [beats/min]], PR (110≤PR≤219 [ms]), QRS (QRS<110 [ms]), QT, QTcF (QTcF for Male<460 and for Female<470 [ms]), or overall interpretation.
Physical examination | Through 365 days
  A full best practice physical examination will be performed by the PI
Clinical Laboratory Tests | Through 365 days
  Measurements of clinical laboratory abnormalities

SECONDARY OUTCOMES:
Evaluation of immunogenicity using a humoral immune function ELISA assay from serum | Through 365 days
  Immunogenicity is measured as having generated anti-HPV type16 L2 and HPV type 31 L2 antibodies after vaccination. The antibody response is measured as a titer.
Evaluation of HPV-Neutralizing Antibodies using an in vitro Pseudovirion-Based HPV-Neutralization Assay (PBNA) | Through 365 days
  Neutralization is measured as having induced anti-HPV antibodies able to protect/neutralize HPV infection in vitro. The neutralization antibody titers are presented as the IC50 titer.

CONTACTS AND LOCATIONS:
Overall Officials: John Nieland, Study Chair — 2A Pharma AB; David Bell, Principal Investigator — Celerion, CRO
Locations (1):
- Celerion Inc., Belfast, Co.Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No